CLINICAL TRIAL: NCT04908436
Title: Investigation of Pharmacokinetics, Safety, and Tolerability of BAY 94-8862 in Male and Female Subjects With Renal Impairment and in Age- and Weight-matched Healthy Subjects Following a Single Oral Dose of 10 mg BAY 94-8862 IR Tablet in a Single-center, Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: A Study to Learn How BAY94-8862 Moves Into, Through and Out of the Body, How Safe it is and How it Affects the Body in Adult Participants With Reduced Kidney Function and in Healthy Participants With Similar Age, Weight and Gender Distribution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14509; 2010-022321-16 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Worsening Chronic Heart Failure; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal renal function (Experimental): Healthy participants with creatinine clearance (CLCR) >80 mL/min received single oral dose of 10 mg BAY94-8862 as an IR tablet under fasting conditions.
  Interventions: Drug: Finerenone (BAY94-8862)
- Mild renal impairment (Experimental): Participants with CLCR 50-80 mL/min received single oral dose of 10 mg BAY94-8862 as an IR tablet under fasting conditions.
  Interventions: Drug: Finerenone (BAY94-8862)
- Moderate renal impairment (Experimental): Participants with CLCR 30-<50 mL/min received single oral dose of 10 mg BAY94-8862 as an IR tablet under fasting conditions.
  Interventions: Drug: Finerenone (BAY94-8862)
- Severe renal impairment (Experimental): Participants with CLCR <30 mL/min received single oral dose of 10 mg BAY94-8862 as an IR tablet under fasting conditions.
  Interventions: Drug: Finerenone (BAY94-8862)

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — 10 mg BAY94-8862 immediate release (IR) tablet, administered orally

SUMMARY:
Researchers are looking for a better way to treat people who have worsening of chronic heart failure, a long-term condition where the heart does not pump blood as well as it should.

In this study researchers wanted to learn more about a new substance called finerenone (BAY94-8862).

Finerenone is a substance that blocks the activation of a protein in the body called mineralocorticoid receptor (MR). An increased activation of MR is involved in the development of hypertension, organ damage and worsening of heart failure. Many patients with worsening chronic heart failure also suffer from chronic kidney disease. Chronic kidney disease is a long-term decrease in the kidneys' ability to work properly.

The researchers studied how finerenone moves into, through and out of the body. The researchers also looked at how safe finerenone is and how it affects the body. The main purpose of this study was to help researchers develop recommendations for the amount of the substance (the dosing) to be given to patients with reduced kidney function.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study specific tests or procedures are done;
* Male participants and female participants without childbearing potential (postmenopausal women with 12 month of spontaneous amenorrhea or with 6 month of spontaneous amenorrhea and serum follicle-stimulating hormone (FSH) levels >30 mIU/mL; women with 6 weeks post bilateral ovarectomy, women with bilateral tubal ligation, and women with hysterectomy);
* Age: 18 to 79 years at the first screening examination;
* Race: White;
* Body mass index (BMI): ≥ 18 and ≤ 34 kg / m2;

Participants with renal impairment

* Creatinine clearance (CLCR) ≤ 80 mL/min determined from a 24 hour urine collection interval 2 - 14 days prior to dosing;
* Stable renal disease, ie a serum creatinine value determined at least 3-6 months before the pre-study visit should not vary by more than 20% from the serum creatinine value determined at the pre-study visit;

Healthy participants

- Mean age and body weight in Group 1 (control group, healthy participants) and Groups 2 - 4 should not vary by more than +/- 10 years and +/- 10 kg, respectively.

Exclusion Criteria:

* Participation in another clinical trial during the preceding 3 months for multiple dose studies and 1 month for single-dose studies; (final examination from previous study to first treatment of new study);
* Exclusion periods from other studies or simultaneous participation in other clinical studies;
* Donation of more than 100 mL of blood within 4 weeks before the first study drug administration or more than 500 mL in the preceding 3 months;
* Regular use of following medication during or within the 1 - 2 weeks preceding the study:

  * concomitant administration of other Aldosterone-antagonists (eg. eplerenone or spironolactone), potassium-sparing diuretics, potassium supplements, nonsteroidal anti-inflammatory drugs like ASS (secondary prevention with a dose of 100 mg daily is allowed), indomethacin or ibuprofen
  * concomitant use of cytochrome P450 isoenzyme 3A4 (CYP3A4) inducers (eg St. John´s wort, rifampicin, carbamazepin, phenytoin, phenobarbital, bosentan)
  * concomitant use of weak to moderate CYP3A4 inhibitors (eg erythromycin, quinupristin/dalfopristin, saquinavir, fluconazole, amiodarone, diltiazem, fluvoxamine, verapamil, valproic acid, fluoxetine, grapefruit juice)
  * strong inhibitors of CYP3A4 (eg human immunodeficiency virus (HIV) protease inhibitors like indinavir, nelfinavir, ritonavir, atazanavir, lopinavir, amprenavir and saquinavir; macrolide/ketolide antibiotics like clarithromycin, telithromycin; antimycotic agents like itraconazole and ketoconazole [topical formulations will be allowed]; nefazodone)
  * moderate and strong inhibitors of cytochrome P450 isoenzyme 2C8 (CYP2C8) (eg gemfibrozil, montelukast, trimethoprim, glitazones)
* Women of childbearing potential, pregnant or lactating women;
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV 1+2);
* Serum potassium level ≥ 5.5 mmol/L;
* Serum sodium level ≤ 130 mmol/L;

For participants with renal impairment

* Acute renal failure;
* Acute nephritis;
* Any organ transplant;
* Failure of any other major organ system other than the kidney;
* Diastolic blood pressure (DBP) > 100 mmHg and/or systolic blood pressure (SBP) > 180 mmHg (at the pre-study examination; readings taken at the end of the dosing interval of antihypertensive medication, if any);
* Heart rate below 45 or above 110 BPM at screening visit;
* Hemoglobin < 8 g/dL;
* Serum albumin < 30 g/L;
* Severe cerebrovascular or cardiac disorders, eg myocardial infarction less than 6 months prior to dosing, congestive heart failure of New York Heart Association (NYHA) grade III or IV, decompensated heart failure, severe arrhythmia requiring antiarrhythmic treatment;

For healthy participants

* A history of relevant diseases of vital organs, of the central nervous system or other organs;
* Systolic blood pressure below 100 mmHg or above 145 mmHg;
* Diastolic blood pressure above 95 mmHg;
* Heart rate below 45 or above 95 BPM at screening visit;
* Clinically relevant deviations of the screened laboratory parameters in clinical chemistry, hematology, or urinalysis from reference range;
* Relevant deviation from the normal range in the clinical examination as judged by the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2011-05-05 (Actual); Study Completion 2012-01-27 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration vs time curve from zero to infinity for total (bound and unbound) drug after single dose administration of BAY94-8862 (AUC) | Up to 96 hours post-dose
  AUC for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Maximum total (bound and unbound) drug concentration in plasma after single dose administration of BAY94-8862 (Cmax) | Up to 96 hours post-dose
  Cmax for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
AUC for unbound drug (AUCu) | Up to 96 hours post-dose
  AUCu for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Cmax for unbound drug (Cmax,u) | Up to 96 hours post-dose
  Cmax,u BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
AUC divided by dose per kg body weight (AUCnorm) | Up to 96 hours post-dose
  AUCnorm for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
AUCnorm for unbound drug (AUCu,norm) | Up to 96 hours post-dose
  AUCu, norm for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Cmax divided by dose per body weight (Cmax,norm) | Up to 96 hours post-dose
  Cmax, norm for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Cmax,norm for unbound drug (Cmax,u,norm) | Up to 96 hours post-dose
  Cmax,u,norm for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)

SECONDARY OUTCOMES:
Plasma renin activity (PRA) | Prior to dosing and 12 hours post-dose
  Change from baseline in plasma renin activity
Plasma angiotensin II | Prior to dosing and 12 hours post-dose
  Change from baseline in plasma angiotensin II
Serum aldosterone | Prior to dosing and 12 hours post-dose
  Change from baseline in serum aldosterone
Plasminogen activator inhibitor-1 (PAI-1) | Prior to dosing and 12 hours post-dose
  Change from baseline in PAI-1
Urinary volume | Prior to dosing up to 24 hours post-dose
  Change in volume of urine excreted
Urinary creatinine | Prior to dosing up to 24 hours post-dose
  Change in urine creatinine concentrations
Urinary electrolytes | Prior to dosing up to 24 hours post-dose
  Change in urinary electrolytes
Half-life associated with the terminal slope (t½) | Up to 96 hours post-dose
  t½ for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Fraction unbound (fu) | 1 hour and 6 hours post-dose
  fu for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
AUC divided by dose (AUC/D) | Up to 96 hours post-dose
  AUC/D for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
AUC from time 0 to the last data point (AUC(0-tlast)) | Up to 96 hours post-dose
  AUC(0-tlast) for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Cmax divided by dose (Cmax/D) | Up to 96 hours post-dose
  Cmax/D for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Time to reach Cmax (tmax) | Up to 96 hours post-dose
  Time to reach Cmax (in case of two identical Cmax values, the first tmax was to be used) for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Mean residence time (MRT) | Up to 96 hours post-dose
  MRT for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Total body clearance of drug calculated after extravascular administration (CL/F) | Up to 96 hours post-dose
  CL/F for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Total body clearance of unbound drug from plasma calculated after oral administration (apparent oral unbound clearance) (CLu/F) | Up to 96 hours post-dose
  CLu/F for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Apparent volume of distribution during terminal phase after extravascular administration (Vz/F) | Up to 96 hours post-dose
  Vz/F for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Amount excreted into urine from 0 to 96 h (end of urine sampling) after study drug administration (AE,ur) | Up to 96 hours post-dose
  AE,ur for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Percent amount excreted into urine from 0 to 96 h (end of urine sampling) after study drug administration (%AE,ur) | Up to 96 hours post-dose
  %AE,ur for BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Renal body clearance of drug (CLR) | Up to 96 hours post-dose
  CLR of BAY94-8862 and its metabolites M1 (BAY1040818), M2 (BAY1088089) and M3 (BAY1088090)
Number of participants with adverse events | Approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Heinig R, Kimmeskamp-Kirschbaum N, Halabi A, Lentini S. Pharmacokinetics of the Novel Nonsteroidal Mineralocorticoid Receptor Antagonist Finerenone (BAY 94-8862) in Individuals With Renal Impairment. Clin Pharmacol Drug Dev. 2016 Nov;5(6):488-501. doi: 10.1002/cpdd.263. Epub 2016 Jul 18. PMID 27431783